CLINICAL TRIAL: NCT06942377
Title: Peking University People's Hospital
Brief Title: Calcium Channel Blocker Amlodipine for Endometrial Cancer Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Wang Jianliu, Peking University People's Hospital, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Peking University
Record Dates: First submitted 2025-03-10; First posted 2025-04-24 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-04

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; calcium channel blocker
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Amlodipine

STUDY DESIGN:
Intervention Model Description: Patients with endometrial cancer who met the inclusion criteria were randomly divided into the control group and the experimental group in a 1:1 ratio according to the random numbers generated in advance (no preset position, no specific object).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participant Group (No Intervention): Progesterone regimen (oral medroxyprogesterone acetate tablet 250mg-500mg/ day or mirena +GnRHa 3.75mg subcutaneous injection monthly)
- Amlodipine Intervention (Experimental): Progesterone regimen (oral medroxyprogesterone acetate tablet 250mg-500mg/ day or Mirena +GnRHa3.75mg subcutaneous injection monthly) combined with Amlodipine 5mg/day. If the patient's blood pressure is higher than 140/90mmHg at 5mg/d, the dose of amlodipine can be increased to 10mg/day
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — Progesterone regimen (oral medroxyprogesterone acetate tablet 250mg-500mg/ day or Mirena +GnRHa3.75mg subcutaneous injection monthly) combined with Amlodipine
  Arms: Amlodipine Intervention

SUMMARY:
To explore the treatment efficacy of Progesterone Therapeutic Regimen Plus Amlodipine in patients with early endometrial carcinoma (EEC) for conservative treatment.

DETAILED DESCRIPTION:
After diagnosed of EEC by hysteroscopy, patients meet the study criteria will be enrolled. The age, height, weight, waistline, blood pressure, drug load, basic history of infertility and family cancer will be collected. Blood tests, including calcium, albumin, fasting blood glucose (FBG), fasting insulin (FINS), blood lipids, sex hormone levels, anti-müllerian hormone (AMH) and renal/liver function tests will be performed before treatment to evacuate their basic conditions.

Patients with endometrial cancer who met the inclusion criteria were randomly divided into the control group and the experimental group in a 1:1 ratio according to the random numbers generated in advance. The administration regimen for the two groups was as follows:

Control group: progesterone regimen (oral medroxyprogesterone acetate tablet 250mg-500mg/ day or Mirena +GnRHa 3.75mg subcutaneous injection monthly); Trial group: progesterone regimen (oral medroxyprogesterone acetate tablet 250mg-500mg/ day or Mirena +GnRHa3.75mg subcutaneous injection monthly) combined with Amlodipine (oral Amlodipine 5mg/ day); The specific selection of progesterone regimen was based on whether the patients had oral progesterone contraindications and if BMI≥28kg/m2 was not suitable for oral progesterone, Mirena +GnRHa regimen was selected. The choice of Amlodipine is based on the results that Amlodipine can inhibite growth in several endometrial cancer cells, PDX model and patient-derived cells.

For patients remained SD after 9 months of treatment but refused hysterectomy, a multiple disciplinary discussion would be held for individual case, and alternative treatment would be given. Maintenance treatment will be recommended for patients with CR, and participants will be followed up for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of endometrial adenocarcinoma G1-2 of the endometrium
2. If the pathology is endometrial cancer, MRI or ultrasound confirms that the lesion is limited to the endometrium or invading the muscle<1/2, that is, FIGO (2009) stage IA
3. Age ≤ 45 years old
4. Require those who wish to retain their reproductive function to sign informed consent
5. No serious internal medicine complications (severe liver and kidney dysfunction)
6. No contraindications for progesterone treatment or pregnancy
7. Has not experienced hypotension more than three times in the past six months and can be regularly monitored for blood pressure
8. Imaging shows no evidence of distant metastasis
9. A. Initial treatment patients: have not used any protective treatment drugs (progestogens, GNRH-a); B. One course of treatment (12 weeks) with incomplete remission of the lesion (partial remission, persistent or progressive lesion); C. Two courses of treatment (24 weeks) with incomplete remission (partial remission, persistent or progressive lesions);

Exclusion Criteria:

1. Tumor invasion of muscle layer>1/2, FIGO (2009) stage IB or above
2. Tumor differentiation into G3 or non endometrioid adenocarcinoma
3. Merge malignant tumors from other parts
4. Individuals with contraindications to conservative treatment or medication use
5. Patients known to have experienced hypotension
6. Patients who have taken other types of antihypertensive drugs regularly in the past

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological cumulative complete response rate after 6 months treatment | Day 1:take medication orally every day；Every three months, undergo hysteroscopy to obtain endometrium for HE and IHC of ER/PR; assessed up to 6-7 months
  No endometrioid carcinoma or any proliferative lesion is found by pathology; imaging examination shows no evidence of a tumor

SECONDARY OUTCOMES:
Recurrence rate | Day 1:take medication orally every day；Every three months, undergo hysteroscopy to obtain endometrium for HE and IHC of ER/PR; up to 12 months after the end of treatment.
  After complete remission, there is evidence of recurrence in pathology, and the imaging examination shows that the lesion recurrences.
Pathological cumulative complete response rate after 12 months treatment | assessed up to 12 months
  The ratio of woman achieved CR after 12 months treatment
Pregnancy rate | Day 1:take medication orally every day；Every three months, undergo hysteroscopy to obtain endometrium for HE and IHC of ER/PR; Through study completion, an average of 1 year
  A pregnancy test shows pregnancy after CR.
Pathological biomarker | Day 1:take medication orally every day；Every three months, undergo hysteroscopy to obtain endometrium for HE and IHC of ER/PR; Through study completion, an average of 1 year
  pathological markers(such as Ki-67, estrogen receptor, progesterone receptor, p53, PTEN, MLH1, PMS2, MSH2, and MSH6) at each hysteroscopy
Adverse reactions | Day 1:take medication orally every day；Every three months, serological testing confirms the effects of drugs on the liver and kidneys; Through study completion, an average of 1 year
  Any unfavorable response resulting from the administration of any pharmaceutical agent utilized as part of the therapeutic regimen.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No